CLINICAL TRIAL: NCT01510431
Title: An Open-label Compassionate Treatment Protocol to Evaluate the Safety and Treatment Outcomes of PROCHYMAL® (Remestemcel-L) Intravenous Infusion in Subjects With Treatment-resistant Crohn's Disease
Brief Title: Safety and Treatment Outcome Study of PROCHYMAL® (Remestemcel-L) Intravenous Infusion in Subjects With Treatment-resistant Crohn's Disease
Status: No longer available | Type: Expanded Access
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Other Study IDs: CRD 620
Record Dates: First submitted 2012-01-09; First posted 2012-01-16 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — remestemcel-l

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: PROCHYMAL (remestemcel-L) — intravenous administration of 200 million cells on days 0, 3, 7, and 14, and then, at investigator discretion, periodically thereafter

SUMMARY:
Protocol 620 provides PROCHYMAL(R) adult human mesenchymal cells to specifically chosen Crohn's disease patients at participating centers who typically have already demonstrated good response in another PROCHYMAL study, are not eligible for other PROCHYMAL studies, and in the view of the investigator, would not benefit significantly from other Crohn's therapies but would benefit from use of PROCHYMAL.

The study is not placebo-controlled or randomized.

ELIGIBILITY:
Inclusion Criteria:

* currently active moderate-to-severe Crohn's disease
* exhausted standard-of-care options
* age 18 to 70 inclusive
* body weight between 30 and 150 kg
* adequate renal function
* not at risk for tuberculosis (TB) activation or re-activation

Exclusion Criteria:

* biologic therapy for Crohn's within last 8 weeks
* confirmed adverse reactions during prior PROCHYMAL study participation
* alcohol or substance abuse, current or within past 6 months
* active HIV or hepatitis B or C infection
* surgery or trauma with 6 weeks
* allergy to bovine or porcine products
* elevated serum liver enzymes
* elevated serum bilirubin
* active malignancy within 5 years (other than some resected skin cancers)
* bacteremia or other serious bacterial or fungal infection within 3 months
* colonic dysplasia
* unstable arrhythmia or serious heart condition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mahboob Rahman, MD, Study Director — Mesoblast, Inc.
Locations (4):
- United States (4):
  - Unviersity of California, San Francisco, San Francisco, California
  - Stormont-Vail, Topeka, Kansas
  - Mount Sinai Hospital, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee